CLINICAL TRIAL: NCT06956079
Title: Effect of End-inspiratory Pause on Gas Exchange During Mediastinal Mass Excision With CO2 Insufflation and One-lung Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4-2025-0232
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Mediastinal Mass Requiring Video-assisted Surgical Excision

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIP-first group (Experimental): EIP is applied for 20 minutes immediately after the initiation of one-lung ventilation, followed by conventional mechanical ventilation.
  Interventions: Procedure: EIP-first
- EIP-later group (Active Comparator): Conventional mechanical ventilation is applied for 20 minutes after the initiation of one-lung ventilation, followed by EIP application.
  Interventions: Procedure: EIP-later

INTERVENTIONS:
Procedure: EIP-first — EIP is applied for 20 minutes immediately after the initiation of one-lung ventilation, followed by conventional mechanical ventilation.
  Arms: EIP-first group
Procedure: EIP-later — Conventional mechanical ventilation is applied for 20 minutes after the initiation of one-lung ventilation, followed by EIP application.
  Arms: EIP-later group

SUMMARY:
" Mediastinal mass excision is typically performed via video-assisted thoracoscopic surgery (VATS). To secure a clear surgical field, the ipsilateral lung must be deflated, achieved through one-lung ventilation (OLV) and intrathoracic CO₂ insufflation. However, OLV increases intrapulmonary shunt due to continued perfusion of the non-ventilated lung, potentially leading to hypoxemia and hypercapnia.

When performed in the supine position, gas exchange becomes more challenging compared to lateral decubitus due to limited gravitational redistribution of blood flow. Although CO₂ insufflation aids surgical exposure through passive lung deflation, it may also increase CVP and PCWP, reduce cardiac output, and raise PaCO₂, contributing to respiratory acidosis.

End-inspiratory pause (EIP), a ventilatory setting that pauses airflow at end-inspiration, prolongs alveolar gas exchange and improves ventilation-perfusion matching. Prior studies show EIP can enhance gas exchange, reduce microatelectasis, and improve CO₂ clearance in patients with acute lung injury. We therefore aimed to assess the effect of EIP application during VATS mediastinal mass excicion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20 to 80 years scheduled for video-assisted thoracoscopic mediastinal tumor resection.
* American Society of Anesthesiologists (ASA) physical status classification of II (patients with mild systemic disease) or III (patients with severe systemic disease limiting activity).

Exclusion Criteria:

* Moderate to severe chronic obstructive pulmonary disease (COPD) according to GOLD criteria: defined as FEV₁/FVC < 0.7 and FEV₁ ≤ 80% of predicted on pulmonary function testing.
* Diffusion capacity of the lung for carbon monoxide (DLCO) < 80% of predicted.
* History of pneumothorax or presence of bullae or blebs on preoperative imaging.
* Inability to read or understand the subject information sheet and consent form.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
PaCO₂ at 20 minutes after each ventilation method | PaCO₂ is assessed at 20 minutes after each ventilation method
  The study aimed to evaluate whether the application of EIP resulted in a significant intergroup difference in PaCO₂.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No